CLINICAL TRIAL: NCT02129205
Title: A PHASE 1 DOSE ESCALATION STUDY EVALUATING THE SAFETY AND TOLERABILITY OF PF-06650808 IN PATIENTS WITH ADVANCED SOLID TUMORS
Brief Title: A Dose Escalation Study of PF-06650808 in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated due to a change in sponsor prioritization.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: B7501001
Record Dates: First submitted 2014-04-30; First posted 2014-05-02 (Estimated); Results first posted 2019-03-29 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2018-12

CONDITIONS: Neoplasms; Breast Cancer
Keywords: solid tumors; triple negative breast cancer; PF-06650808; Phase 1
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — PF-06650808

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PF-06650808 (Experimental)
  Interventions: Drug: PF-06650808

INTERVENTIONS:
Drug: PF-06650808 — Dose Escalation Phase [Part 1] - PF-06650808 will be administered at doses starting at 0.2 mg/kg. Increases in dose will continue until MTD is determined.
Drug: PF-06650808 — Dose Expansion Phase [Part 2] - Patients will be treated at the MTD or Recommended Phase 2 dose selected in Part 1.

SUMMARY:
To assess the safety and tolerability at increasing dose levels of PF-06650808 in patients with advanced solid tumors in order to determine the maximum tolerated dose and select the recommended Phase 2 dose.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced/metastatic solid tumor that is resistant to standard therapy or for which no standard therapy is available
* Previously treated metastatic triple negative breast cancer that expresses Notch3 with at least one measurable lesion
* Adequate bone marrow, renal and liver function

Exclusion Criteria:

* Major surgery, radiation therapy or systemic anti-cancer therapy within 4 weeks of starting study treatment
* Patients with known symptomatic brain metastases requiring steroids
* Prior treatment with a compound of the same mechanism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (11):
- United States (11):
  - Ronald Reagan UCLA Medical Center, Drug Information Center, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA Hematology/Oncology, Los Angeles, California
  - Westwood Bowyer Clinic, Los Angeles, California
  - Santa Monica - UCLA Medical Center & Orthopaedic Hospital, Santa Monica, California
  - UCLA Hematology/Oncology - Santa Monica, Santa Monica, California
  - The Ohio State University James Cancer Hospital, Columbus, Ohio
  - The OSU Investigational Drug Services, Columbus, Ohio
  - The OSU Stephanie Spielman Comprehensive Breast Center, Columbus, Ohio
  - The Ohio State University Martha Morehouse Medical Plaza, Columbus, Ohio
  - South Texas Accelerated Research Therapeutics, LLC (START), San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Rosen LS, Wesolowski R, Baffa R, Liao KH, Hua SY, Gibson BL, Pirie-Shepherd S, Tolcher AW. A phase I, dose-escalation study of PF-06650808, an anti-Notch3 antibody-drug conjugate, in patients with breast cancer and other advanced solid tumors. Invest New Drugs. 2020 Feb;38(1):120-130. doi: 10.1007/s10637-019-00754-y. Epub 2019 Mar 18. PMID 30887250
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7501001&StudyName=A%20Dose%20Escalation%20Study%20of%20PF-06650808%20in%20Patients%20with%20Advanced%20Solid%20Tumors%20

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-06650808 0.2 mg/kg (Part 1): PF-06650808 0.2 mg/kg was administered intravenously on Day 1 of each 21-day cycle for 4 months or until disease progression, participant refusal or unacceptable toxicity occurred.
- PF-06650808 0.4 mg/kg (Part 1): PF-06650808 0.4 mg/kg was administered intravenously on Day 1 of each 21-day cycle for 4 months or until disease progression, participant refusal or unacceptable toxicity occurred.
- PF-06650808 0.8 mg/kg (Part 1): PF-06650808 0.8 mg/kg was administered intravenously on Day 1 of each 21-day cycle for 4 months or until disease progression, participant refusal or unacceptable toxicity occurred.
- PF-06650808 1.6 mg/kg (Part 1): PF-06650808 1.6 mg/kg was administered intravenously on Day 1 of each 21-day cycle for 4 months or until disease progression, participant refusal or unacceptable toxicity occurred.
- PF-06650808 2.0 mg/kg (Part 1): PF-06650808 2.0 mg/kg was administered intravenously on Day 1 of each 21-day cycle for 4 months or until disease progression, participant refusal or unacceptable toxicity occurred.
- PF-06650808 2.4 mg/kg (Part 1): PF-06650808 2.4 mg/kg was administered intravenously on Day 1 of each 21-day cycle for 4 months or until disease progression, participant refusal or unacceptable toxicity occurred.
- PF-06650808 3.0 mg/kg (Part 1): PF-06650808 3.0 mg/kg was administered intravenously on Day 1 of each 21-day cycle for 4 months or until disease progression, participant refusal or unacceptable toxicity occurred.
- PF-06650808 3.6 mg/kg (Part 1): PF-06650808 3.6 mg/kg was administered intravenously on Day 1 of each 21-day cycle for 4 months or until disease progression, participant refusal or unacceptable toxicity occurred.
- PF-06650808 4.68 mg/kg (Part 1): PF-06650808 4.68 mg/kg was administered intravenously on Day 1 of each 21-day cycle for 4 months or until disease progression, participant refusal or unacceptable toxicity occurred.
- PF-06650808 2.4mg/kg (Part 2): Part 2 of PF-06650808 was planned to inlcude the participants with Notch3 expressing triple negative breast cancer at the maximum tolerated dose (MTD). The MTD of PF-06650808 was determined to be 2.4 mg/kg in Part 1. The Part 2 was not conducted as the termination of study.
Period: Overall Study
Arm/Group | PF-06650808 0.2 mg/kg (Part 1) | PF-06650808 0.4 mg/kg (Part 1) | PF-06650808 0.8 mg/kg (Part 1) | PF-06650808 1.6 mg/kg (Part 1) | PF-06650808 2.0 mg/kg (Part 1) | PF-06650808 2.4 mg/kg (Part 1) | PF-06650808 3.0 mg/kg (Part 1) | PF-06650808 3.6 mg/kg (Part 1) | PF-06650808 4.68 mg/kg (Part 1) | PF-06650808 2.4mg/kg (Part 2)
Started | 2 | 2 | 2 | 2 | 7 | 11 | 6 | 6 | 2 | 0
Completed | 1 | 2 | 2 | 2 | 4 | 7 | 2 | 4 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 3 | 4 | 4 | 2 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0
Not completed — Other | 1 | 0 | 0 | 0 | 2 | 3 | 3 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants who received at least 1 dose of study treatment.
Groups:
- PF-06650808 2.4 mg/kg (Part 2): Part 2 of PF-06650808 was planned to inlcude the participants with Notch3 expressing triple negative breast cancer at the MTD. The MTD of PF-06650808 was determined to be 2.4 mg/kg in Part 1. The Part 2 was not conducted as the termination of study.
- Total: Total of all reporting groups
Arm/Group | PF-06650808 0.2 mg/kg (Part 1) | PF-06650808 0.4 mg/kg (Part 1) | PF-06650808 0.8 mg/kg (Part 1) | PF-06650808 1.6 mg/kg (Part 1) | PF-06650808 2.0 mg/kg (Part 1) | PF-06650808 2.4 mg/kg (Part 1) | PF-06650808 3.0 mg/kg (Part 1) | PF-06650808 3.6 mg/kg (Part 1) | PF-06650808 4.68 mg/kg (Part 1) | PF-06650808 2.4 mg/kg (Part 2) | Total
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 7 | 11 | 6 | 6 | 2 | 0 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (6.4) | 69.5 (3.5) | 55 (24) | 49.5 (2.1) | 51.9 (14.7) | 59.9 (9.8) | 59.3 (13.8) | 60.8 (4.7) | 42 (28.3) |  | 57.2 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 1 | 7 | 11 | 3 | 6 | 2 | 0 | 35
  Male | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 5
Race/Ethnicity, Customized [Number; unit: participants]
  White | 2 | 1 | 2 | 2 | 6 | 8 | 5 | 4 | 2 |  | 32
  Black | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 |  | 4
  Asian | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 |  | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLT) (Part 1)
Description: Severity of AEs (adverse events ) was graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. For the purpose of dose escalation, any of the following AEs which were not considered related to disease progression occurring in the first cycle of treatment (21 days) were classified as DLTs: 1) Hematologic: Grade 4 neutropenia lasting >7 days; Febrile neutropenia; Grade>=3 neutropenia with infection; Any grade thrombocytopenia associated with clinically significant or life threatening bleeding; Grade 4 thrombocytopenia >=72 hours or platelets<=10,000/mm3 regardless of duration. 2) Non hematologic: Grade>=3 toxicities except those that had not been maximally treated; Delayed by more than 2 weeks in receiving the next scheduled cycle due to persisting toxicities not attributable to disease progression. 3) clinically important or persistent toxicities may have been considered a DLT following review by the Sponsor and the investigators.
Time Frame: Day 1 up to Day 21
Population: The safety analysis set was used, which included all enrolled participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06650808 0.2 mg/kg (Part 1) | PF-06650808 0.4 mg/kg (Part 1) | PF-06650808 0.8 mg/kg (Part 1) | PF-06650808 1.6 mg/kg (Part 1) | PF-06650808 2.0 mg/kg (Part 1) | PF-06650808 2.4 mg/kg (Part 1) | PF-06650808 3.0 mg/kg (Part 1) | PF-06650808 3.6 mg/kg (Part 1) | PF-06650808 4.68 mg/kg (Part 1)
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 7 | 11 | 6 | 6 | 2
Participants
  Yes | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 2
  No | 2 | 2 | 2 | 2 | 7 | 8 | 4 | 5 | 0

2. Primary Outcome: Percentage of Participants With Objective Response (Part 1 and Part 2)
Description: Assessment of response was made using Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. A participant achieved complete response (CR) if both target and non-target lesions achieved CR, no new lesions; achieved partial response (PR) if target lesions achieved CR or PR, non-target lesions were assessed as non-CR/non-PD (progressive disease), indeterminate or missing, and no new lesions. For target lesions, CR: complete disappearance of all target lesions except nodal disease (target nodes must decrease to normal size); PR: >= 30% decrease under baseline of the sum of diameters of all target measurable lesions. For non-target lesions, CR: disappearance of all non-target lesions and normalization of tumor marker levels and all lymph nodes must be normal in size; non-CR/non-PD: persistence of any non-target lesions and/or tumor marker level above the normal limits. The overall objective response was defined as confirmed CR and PR.
Time Frame: Day 1 and every 6 weeks until disease progression, unacceptable toxicity, or up to 3 years
Population: The analysis population included all participants who received at least 1 dose of study medication and had both baseline and at least 1 post-baseline tumor assessments. The study was prematurely terminated prior to the start of dose expansion phase (Part 2).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PF-06650808 0.2 mg/kg (Part 1) | PF-06650808 0.4 mg/kg (Part 1) | PF-06650808 0.8 mg/kg (Part 1) | PF-06650808 1.6 mg/kg (Part 1) | PF-06650808 2.0 mg/kg (Part 1) | PF-06650808 2.4 mg/kg (Part 1) | PF-06650808 3.0 mg/kg (Part 1) | PF-06650808 3.6 mg/kg (Part 1) | PF-06650808 4.68 mg/kg (Part 1) | PF-06650808 2.4 mg/kg (Part 2)
Number analyzed (Participants) | 2 | 2 | 1 | 2 | 6 | 7 | 4 | 5 | 2 | 0
Percentage of participants | 0 [0.0 to 84.2] | 0 [0.0 to 84.2] | 0 [0.0 to 97.5] | 0 [0.0 to 84.2] | 16.7 [0.4 to 64.1] | 14.3 [0.4 to 57.9] | 0 [0.0 to 60.2] | 20.0 [0.5 to 71.6] | 0 [0.0 to 84.2] |

3. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) (Part 1 and Part 2)
Description: AE was defined as any untoward medical occurrence in a clinical investigation participant administered a product or medical device, regardless of the causal relationship to study treatment. Treatment-emergent AEs (TEAEs) were defined as AEs which occurred for the first time during the effective duration of treatment or AEs that increased in severity during treatment. Serious AEs (SAEs) were defined as any untoward medical occurrence at any dose that resulted in death; was life-threatening (immediate risk of death); required inpatient hospitalization or caused prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduction normal life functions). AEs included SAEs and non-serious AEs. Causality to study treatment was determined by the investigator. Severity was graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: 3 years
Population: The safety analysis set was used, which included all enrolled participants who received at least one dose of study medication. The study was prematurely terminated prior to the start of dose expansion phase (Part 2).
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06650808 0.2 mg/kg (Part 1) | PF-06650808 0.4 mg/kg (Part 1) | PF-06650808 0.8 mg/kg (Part 1) | PF-06650808 1.6 mg/kg (Part 1) | PF-06650808 2.0 mg/kg (Part 1) | PF-06650808 2.4 mg/kg (Part 1) | PF-06650808 3.0 mg/kg (Part 1) | PF-06650808 3.6 mg/kg (Part 1) | PF-06650808 4.68 mg/kg (Part 1) | PF-06650808 2.4 mg/kg (Part 2)
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 7 | 11 | 6 | 6 | 2 | 0
Participants
  All causalities AE Grade 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 |
  All causalities AE Grade 2 | 2 | 1 | 1 | 2 | 1 | 2 | 1 | 1 | 0 |
  All causalities AE Grade 3 | 0 | 1 | 0 | 0 | 5 | 8 | 2 | 4 | 1 |
  All causalities AE Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 |
  All causalities AE Grade 5 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 |
  All causalities SAE Grade 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 |
  All causalities SAE Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  All causalities SAE Grade 3 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 1 |
  All causalities SAE Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 |
  All causalities SAE Grade 5 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 |
  Treatment related AE Grade 1 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 |
  Treatment related AE Grade 2 | 0 | 0 | 0 | 1 | 2 | 4 | 1 | 1 | 0 |
  Treatment related AE Grade 3 | 0 | 0 | 0 | 0 | 4 | 6 | 3 | 4 | 1 |
  Treatment related AE Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 |
  Treatment related AE Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Treatment related SAE Grade 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Treatment related SAE Grade 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 |
  Treatment related SAE Grade 3 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 |
  Treatment related SAE Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 |
  Treatment related SAE Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |

4. Secondary Outcome: Number of Participants With Laboratory Abnormalities Without Regard to Baseline (Hematology) (Part 1 and Part 2)
Description: Hematology evaluation included hemoglobin, platelets, white blood cell, absolute neutrophils, absolute lymphocytes, absolute monocytes, absolute eosinophils and absolute basophils. The participants who experienced laboratory test abnormalities were determined by investigators.
Time Frame: 3 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06650808 0.2 mg/kg (Part 1) | PF-06650808 0.4 mg/kg (Part 1) | PF-06650808 0.8 mg/kg (Part 1) | PF-06650808 1.6 mg/kg (Part 1) | PF-06650808 2.0 mg/kg (Part 1) | PF-06650808 2.4 mg/kg (Part 1) | PF-06650808 3.0 mg/kg (Part 1) | PF-06650808 3.6 mg/kg (Part 1) | PF-06650808 4.68 mg/kg (Part 1) | PF-06650808 2.4 mg/kg (Part 2)
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 7 | 11 | 6 | 6 | 2 | 0
Participants
  Anemia | 1 | 2 | 2 | 1 | 4 | 6 | 5 | 3 | 2 |
  Hemoglobin increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Lymphocyte count increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Lymphopenia | 2 | 1 | 2 | 1 | 4 | 9 | 4 | 4 | 2 |
  Neutrophils count decreased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Patelets count decreased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  White blood cells decreased | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 0 | 0 |

5. Secondary Outcome: Number of Participants With Laboratory Abnormalities Without Regard to Baseline (Chemistries) (Part 1 and Part 2)
Description: Chemistry evaluation included alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, sodium, potassium, magnesium, chloride, calcium, total bilirubin, blood urea nitrogen (BUN) or urea, creatinine, uric acid, glucose (non-fasted), albumin, phosphorus, bicarbonate or carbon dioxide, total protein and lactate dehydrogenase. The participants who experienced laboratory test abnormalities were determined by investigators.
Time Frame: 3 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06650808 0.2 mg/kg (Part 1) | PF-06650808 0.4 mg/kg (Part 1) | PF-06650808 0.8 mg/kg (Part 1) | PF-06650808 1.6 mg/kg (Part 1) | PF-06650808 2.0 mg/kg (Part 1) | PF-06650808 2.4 mg/kg (Part 1) | PF-06650808 3.0 mg/kg (Part 1) | PF-06650808 3.6 mg/kg (Part 1) | PF-06650808 4.68 mg/kg (Part 1) | PF-06650808 2.4 mg/kg (Part 2)
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 7 | 11 | 6 | 6 | 2 | 0
Participants
  Alanine aminotransferase (ALT) increased | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 1 |
  Alkaline phosphatase increased | 1 | 0 | 1 | 1 | 4 | 3 | 2 | 1 | 1 |
  Aspartate aminotransferase (AST) increased | 0 | 1 | 1 | 0 | 4 | 4 | 0 | 1 | 1 |
  Bilirubin (Total) increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Creatinine increased | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 |
  Hypercalcemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Hyperglycemia | 0 | 1 | 1 | 2 | 2 | 4 | 5 | 3 | 0 |
  Hyperkalemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Hypermagnesemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Hypernatremia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Hypoalbuminemia | 0 | 0 | 0 | 0 | 1 | 4 | 2 | 1 | 1 |
  Hypocalcemia | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 |
  Hypoglycemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Hypokalemia | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 |
  Hypomagnesemia | 1 | 0 | 1 | 0 | 2 | 2 | 3 | 0 | 1 |
  Hyponatremia | 1 | 1 | 0 | 0 | 2 | 3 | 1 | 2 | 0 |
  Hypophosphatemia | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 |

6. Secondary Outcome: Number of Participants With Laboratory Abnormalities Without Regard to Baseline (Urinalysis) (Part 1 and Part 2)
Description: Urinalysis included urine protein. Microscopic analyses were performed if dipstick was abnormal. The participants who experienced laboratory test abnormalities were determined by investigators.
Time Frame: 3 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06650808 0.2 mg/kg (Part 1) | PF-06650808 0.4 mg/kg (Part 1) | PF-06650808 0.8 mg/kg (Part 1) | PF-06650808 1.6 mg/kg (Part 1) | PF-06650808 2.0 mg/kg (Part 1) | PF-06650808 2.4 mg/kg (Part 1) | PF-06650808 3.0 mg/kg (Part 1) | PF-06650808 3.6 mg/kg (Part 1) | PF-06650808 4.68 mg/kg (Part 1) | PF-06650808 2.4 mg/kg (Part 2)
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 6 | 10 | 5 | 6 | 1 | 0
Participants | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |

7. Secondary Outcome: Number of Participants With Vital Signs Meeting Categorical Summarization Criteria (Part 1 and Part 2)
Description: Vital Signs tests included systolic and diastolic blood pressure (BP) and pulse rate of seated supine and standing . Vital signs categorical summarization criteria were 1), supine and standing BP: systolic (SBP) greater than or equal to (>=) 30 millimeters of mercury (mm Hg) change from baseline, systolic less than (<) 90 mm Hg; diastolic BP (DBP) >=20 mm Hg change from baseline, diastolic <50 mm Hg; 2), supine and standing pulse rate <40 or greater than (>) 120 beats per minute (bpm).
Time Frame: 3 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06650808 0.2 mg/kg (Part 1) | PF-06650808 0.4 mg/kg (Part 1) | PF-06650808 0.8 mg/kg (Part 1) | PF-06650808 1.6 mg/kg (Part 1) | PF-06650808 2.0 mg/kg (Part 1) | PF-06650808 2.4 mg/kg (Part 1) | PF-06650808 3.0 mg/kg (Part 1) | PF-06650808 3.6 mg/kg (Part 1) | PF-06650808 4.68 mg/kg (Part 1) | PF-06650808 2.4 mg/kg (Part 2)
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 7 | 9 | 6 | 6 | 2 | 0
Participants
  Sitting Systolic BP < 90 mmHg | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 |
  Sitting Diastolic BP < 50 mmHg | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 |
  Sitting Pulse Rate < 40 BPM | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Sitting Pulse Rate > 120 BPM | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 0 |
  Supine Systolic BP < 90: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Supine Systolic BP < 90 |  |  |  |  |  | 0 |  |  |  |
  Supine Diastolic BP < 50 mmHg: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Supine Diastolic BP < 50 mmHg |  |  |  |  |  | 0 |  |  |  |
  Supine Pulse Rate < 40 BPM: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Supine Pulse Rate < 40 BPM |  |  |  |  |  | 0 |  |  |  |
  Supine Pulse Rate > 120 BPM: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Supine Pulse Rate > 120 BPM |  |  |  |  |  | 0 |  |  |  |
  Systolic BP < 90 mmHg: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0
  Systolic BP < 90 mmHg |  |  |  |  |  | 1 | 0 |  |  |
  Diastolic BP < 50 mmHg: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0
  Diastolic BP < 50 mmHg |  |  |  |  |  | 1 | 0 |  |  |
  Pulse Rate < 40 BPM: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0
  Pulse Rate < 40 BPM |  |  |  |  |  | 0 | 0 |  |  |
  Pulse Rate > 120 BPM: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0
  Pulse Rate > 120 BPM |  |  |  |  |  | 0 | 0 |  |  |
  Increase: Sitting Systolic BP >= 30 mmHg: number analyzed (Participants) | 2 | 2 | 2 | 2 | 7 | 8 | 6 | 6 | 2 | 0
  Increase: Sitting Systolic BP >= 30 mmHg | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 |
  Increase: Sitting Diastolic BP >= 20 mmHg: number analyzed (Participants) | 2 | 2 | 2 | 2 | 7 | 8 | 6 | 6 | 2 | 0
  Increase: Sitting Diastolic BP >= 20 mmHg | 0 | 0 | 1 | 0 | 1 | 3 | 2 | 4 | 0 |
  Increase: Systolic BP >= 30 mmHg: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
  Increase: Systolic BP >= 30 mmHg |  |  |  |  |  | 0 |  |  |  |
  Increase: Diastolic BP >= 20 mmHg: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
  Increase: Diastolic BP >= 20 mmHg |  |  |  |  |  | 0 |  |  |  |
  Decrease: Sitting Systolic BP >= 30 mmHg: number analyzed (Participants) | 2 | 2 | 2 | 2 | 7 | 8 | 6 | 6 | 2 | 0
  Decrease: Sitting Systolic BP >= 30 mmHg | 0 | 1 | 0 | 0 | 2 | 1 | 2 | 1 | 0 |
  Decrease: Sitting Diastolic BP >= 20 mmHg: number analyzed (Participants) | 2 | 2 | 2 | 2 | 7 | 8 | 6 | 6 | 2 | 0
  Decrease: Sitting Diastolic BP >= 20 mmHg | 0 | 1 | 1 | 0 | 2 | 2 | 0 | 1 | 0 |
  Decrease: Systolic BP >= 30 mmHg: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
  Decrease: Systolic BP >= 30 mmHg |  |  |  |  |  | 1 |  |  |  |
  Decrease: Diastolic BP >= 20 mmHg: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
  Decrease: Diastolic BP >= 20 mmHg |  |  |  |  |  | 2 |  |  |  |

8. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) (Part 1 and Part 2)
Description: Maximum observed serum concentration (Cmax) of ADC (PF-06650808), total antibody (PF-06460005) and unconjugated payload (PF-06380101) were observed directly from data. PF-06650808 is comprised of an antibody (PF-06460005) and a cytotoxic agent (PF-06380101).
Time Frame: Pre-dose, 1, 4 and 24 hours post-dose, Days 4, 8 and 15 in Cycle 1 and Cycle 4
Population: The PK parameter analysis population was defined as all enrolled participants treated who had sufficient information to estimate at least 1 of the PK parameters of interest. The study was prematurely terminated prior to the start of dose expansion phase (Part 2).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06650808 0.2 mg/kg (Part 1) | PF-06650808 0.4 mg/kg (Part 1) | PF-06650808 0.8 mg/kg (Part 1) | PF-06650808 1.6 mg/kg (Part 1) | PF-06650808 2.0 mg/kg (Part 1) | PF-06650808 2.4 mg/kg (Part 1) | PF-06650808 3.0 mg/kg (Part 1) | PF-06650808 3.6 mg/kg (Part 1) | PF-06650808 4.68 mg/kg (Part 1) | PF-06650808 2.4 mg/kg (Part 2)
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 7 | 11 | 6 | 6 | 2 | 0
ng/mL
  Serum PF-06650808 (ADC)_Cycle 1 | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 6200 and 4290 ng/mL, respectively. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 11000 and 8030 ng/mL, respectively. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 18100 and 19400 ng/mL, respectively. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values.Individual participant values are 34600 and 34900 ng/mL, respectively. | 59440 (33) | 54220 (29) | 76480 (27) | 71390 (38) | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values.Individual participant values are 141000 and 92200 ng/mL, respectively |
  Serum PF-06460005 (Total Antibody)_Cycle 1 | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values.Individual participant values are 5000 and 3690 ng/mL, respectively. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values.Individual participant values are 8920 and 7860 ng/mL, respectively. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values.Individual participant values are 21600 and 17700 ng/mL, respectively. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 30800 and 26800 ng/mL, respectively. | 48840 (29) | 54120 (17) | 93530 (53) | 65810 (35) | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values.Individual participant values are 99600 and 62400 ng/mL, respectively. |
  Serum PF-06380101 (Unconjugated Payload)_Cycle 1 | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 0.735 and 0.627 ng/mL, respectively. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 1.180 and 0.536 ng/mL, respectively. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 2.530 and 2.900 ng/mL, respectively. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 2.430 and 6.450 ng/mL, respectively. | 6.495 (75) | 5.916 (81) | 10.680 (30) | 9.060 (82) | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 26.100 and 14.400 ng/mL, respectively. |
  Serum PF-06650808 (ADC)_Cycle 4: number analyzed (Participants) | 0 | 1 | 1 | 2 | 4 | 4 | 0 | 2 | 0 | 0
  Serum PF-06650808 (ADC)_Cycle 4 |  | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values is 11400 ng/mL. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values is 18200 ng/mL. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 36700 and 38100 ng/mL, respectively. | 46240 (12) | 43910 (17) |  | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 36100 and 64900 ng/mL, respectively. |  |
  Serum PF-06460005 (Total Antibody)_Cycle 4: number analyzed (Participants) | 0 | 1 | 1 | 2 | 4 | 4 | 0 | 2 | 0 | 0
  Serum PF-06460005 (Total Antibody)_Cycle 4 |  | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values is 9920 ng/mL. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values is 11900 ng/mL. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 35100 and 51500 ng/mL, respectively. | 41610 (34) | 50640 (23) |  | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 62400 and 108000 ng/mL, respectively. |  |
  Serum PF-06380101 (Unconjugated Payload)_Cycle 4: number analyzed (Participants) | 0 | 1 | 1 | 2 | 4 | 4 | 0 | 2 | 0 | 0
  Serum PF-06380101 (Unconjugated Payload)_Cycle 4 |  | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values is 1.200 ng/mL. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values is 2.180 ng/mL. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 2.220 and 4.730 ng/mL, respectively. | 4.518 (78) | 4.081 (54) |  | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 2.800 and 15.700 ng/mL, respectively. |  |

9. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) (Part 1 and Part 2)
Description: Tmax of ADC (PF-06650808), total antibody (PF-06460005) and unconjugated payload (PF-06380101) were observed directly from data as time of first occurrence.
Time Frame: Pre-dose, 1, 4 and 24 hours post-dose, Days 4, 8 and 15 in Cycle 1 and Cycle 4
Population: as for outcome 8
Measure: Median (Full Range); unit: hr
Arm/Group | PF-06650808 0.2 mg/kg (Part 1) | PF-06650808 0.4 mg/kg (Part 1) | PF-06650808 0.8 mg/kg (Part 1) | PF-06650808 1.6 mg/kg (Part 1) | PF-06650808 2.0 mg/kg (Part 1) | PF-06650808 2.4 mg/kg (Part 1) | PF-06650808 3.0 mg/kg (Part 1) | PF-06650808 3.6 mg/kg (Part 1) | PF-06650808 4.68 mg/kg (Part 1) | PF-06650808 2.4 mg/kg (Part 2)
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 7 | 11 | 6 | 6 | 2 | 0
hr
  Serum PF-06650808 (ADC)_Cycle 1 | 0.967 [0.950 to 0.983] | 0.974 [0.917 to 1.03] | 0.967 [0.967 to 0.967] | 1.01 [0.983 to 1.03] | 0.967 [0.917 to 1.08] | 1.03 [0.933 to 4.05] | 1.06 [0.967 to 4.00] | 1.04 [0.917 to 4.08] | 1.45 [1.15 to 1.75] |
  Serum PF-06460005 (Total Antibody)_Cycle 1 | 0.967 [0.950 to 0.983] | 0.974 [0.917 to 1.03] | 0.967 [0.967 to 0.967] | 1.01 [0.983 to 1.03] | 1.08 [0.917 to 4.02] | 1.02 [0.933 to 3.98] | 1.04 [0.967 to 4.00] | 1.04 [0.950 to 4.08] | 1.45 [1.15 to 1.75] |
  Serum PF-06380101 (Unconjugated Payload)_Cycle 1 | 25.3 [25.2 to 25.4] | 24.6 [23.4 to 25.8] | 48.5 [24.8 to 72.1] | 24.6 [23.8 to 25.4] | 24.0 [22.1 to 71.6] | 24.3 [23.0 to 72.3] | 57.9 [23.1 to 75.9] | 69.1 [22.4 to 73.0] | 47.7 [23.8 to 71.6] |
  Serum PF-06650808 (ADC)_Cycle 4: number analyzed (Participants) | 0 | 1 | 1 | 2 | 4 | 4 | 0 | 2 | 0 | 0
  Serum PF-06650808 (ADC)_Cycle 4 |  | 0.917 [0.917 to 0.917] | 0.917 [0.917 to 0.917] | 1.00 [0.900 to 1.10] | 2.34 [0.933 to 5.00] | 1.03 [0.917 to 1.07] |  | 2.47 [0.933 to 4.00] |  |
  Serum PF-06460005 (Total Antibody)_Cycle 4: number analyzed (Participants) | 0 | 1 | 1 | 2 | 4 | 4 | 0 | 2 | 0 | 0
  Serum PF-06460005 (Total Antibody)_Cycle 4 |  | 0.917 [0.917 to 0.917] | 0.917 [0.917 to 0.917] | 2.55 [1.10 to 4.00] | 1.00 [0.933 to 1.05] | 1.05 [0.917 to 22.1] |  | 0.925 [0.917 to 0.933] |  |
  Serum PF-06380101 (Unconjugated Payload)_Cycle 4: number analyzed (Participants) | 0 | 1 | 1 | 2 | 4 | 4 | 0 | 2 | 0 | 0
  Serum PF-06380101 (Unconjugated Payload)_Cycle 4 |  | 23.4 [23.4 to 23.4] | 24.6 [24.6 to 24.6] | 13.5 [4.00 to 23.0] | 23.5 [21.9 to 25.2] | 46.4 [5.00 to 70.0] |  | 23.6 [23.1 to 24.0] |  |

10. Secondary Outcome: Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) (Part 1 and Part 2)
Description: Tau refers to the dosing interval, and it equals to 504 hours (3 weeks) of ADC (PF-06650808), total antibody (PF-06460005) and unconjugated payload (PF-06380101) were determined using linear/log trapezoidal method.
Time Frame: Pre-dose, 1, 4 and 24 hours post-dose, Days 4, 8 and 15 in Cycle 1 and Cycle 4
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-06650808 0.2 mg/kg (Part 1) | PF-06650808 0.4 mg/kg (Part 1) | PF-06650808 0.8 mg/kg (Part 1) | PF-06650808 1.6 mg/kg (Part 1) | PF-06650808 2.0 mg/kg (Part 1) | PF-06650808 2.4 mg/kg (Part 1) | PF-06650808 3.0 mg/kg (Part 1) | PF-06650808 3.6 mg/kg (Part 1) | PF-06650808 4.68 mg/kg (Part 1) | PF-06650808 2.4 mg/kg (Part 2)
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 6 | 11 | 5 | 5 | 1 | 0
ng*hr/mL
  Serum PF-06650808 (ADC)_Cycle 1 | NA (NA) — Summary statistics were not presented if fewer than 3 partipants had reportable parameter values. Individual participant values are 156000 and 105000 ng.hr/mL, respectively. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 394000 and 255000 ng.hr/mL, respectively. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 515000 and 567000 ng.hr/mL, respectively. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 1290000 and 1070000 ng.hr/mL, respectively. | 1786000 (17) | 2147000 (33) | 3659000 (31) | 2956000 (39) | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values is 4180000 ng.hr/mL. |
  Serum PF-06460005 (Total Antibody)_Cycle 1: number analyzed (Participants) | 1 | 2 | 1 | 2 | 6 | 10 | 5 | 5 | 1 | 0
  Serum PF-06460005 (Total Antibody)_Cycle 1 | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 122000 ng.hr/mL. | NA (NA) — Summary statistics were not presented if fewer than 3 particpants had reportable parameter values. Individual participant values are 371000 and 265000 ng.hr/mL, respectively. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 689000 ng.hr/mL. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 1290000 and 1070000 ng.hr/mL, respectively. | 2385000 (24) | 3078000 (36) | 5116000 (31) | 3571000 (48) | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values is 4270000 ng.hr/mL. |
  Serum PF-06380101 (Unconjugated Payload)_Cycle 1: number analyzed (Participants) | 2 | 1 | 2 | 2 | 6 | 9 | 4 | 5 | 1 | 0
  Serum PF-06380101 (Unconjugated Payload)_Cycle 1 | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 76.300 and 46.600 ng.hr/mL, respectively. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 48.900 ng.hr/mL. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 291.000 and 228.000 ng.hr/mL, respectively. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 300.000 and 576.000 ng.hr/mL, respectively. | 814.700 (96) | 671.500 (103) | 1307.000 (19) | 1082.000 (88) | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 2060.000 ng.hr/mL. |
  Serum PF-06650808 (ADC)_Cycle 4: number analyzed (Participants) | 0 | 1 | 1 | 2 | 4 | 4 | 0 | 2 | 0 | 0
  Serum PF-06650808 (ADC)_Cycle 4 |  | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 365000 ng.hr/mL. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 578000 ng.hr/mL. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participants values are 1550000 and 1150000 ng.hr/mL, respectively. | 1690000 (18) | 1899000 (31) |  | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 1400000 and 2600000 ng.hr/mL, respectively. |  |
  Serum PF-06460005 (Total Antibody)_Cycle 4: number analyzed (Participants) | 0 | 1 | 1 | 2 | 4 | 3 | 0 | 2 | 0 | 0
  Serum PF-06460005 (Total Antibody)_Cycle 4 |  | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 399000 ng.hr/mL. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 593000 ng.hr/mL. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 2130000 and 1720000 ng.hr/mL, respectively. | 2234000 (20) | 2901000 (33) |  | NA (NA) — Summary statistics were not presented if fewer than 3 participants reportable parameter values. Individual participant values are 3160000 and 6060000 ng.hr/mL, respectively. |  |
  Serum PF-06380101 (Unconjugated Payload)_Cycle 4: number analyzed (Participants) | 0 | 1 | 1 | 2 | 4 | 4 | 0 | 2 | 0 | 0
  Serum PF-06380101 (Unconjugated Payload)_Cycle 4 |  | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 113.00 ng.hr/mL. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 186.000 ng.hr/mL. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 304.000 and 403.000 ng.hr/mL, respectively. | 507.400 (90) | 486.600 (78) |  | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 273.000 and 2040.000 ng.hr/mL, respectively. |  |

11. Secondary Outcome: Clearance (CL) (Part 1 and Part 2)
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. CL was calculated as dose/AUCinf, where AUCinf was the area under the serum concentration-time profile from time 0 extrapolated to infinite time. CL was only for PF-06650808 (ADC) and Cycle 1.
Time Frame: Pre-dose, 1, 4 and 24 hours post-dose, Days 4, 8 and 15 in Cycle 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | PF-06650808 0.2 mg/kg (Part 1) | PF-06650808 0.4 mg/kg (Part 1) | PF-06650808 0.8 mg/kg (Part 1) | PF-06650808 1.6 mg/kg (Part 1) | PF-06650808 2.0 mg/kg (Part 1) | PF-06650808 2.4 mg/kg (Part 1) | PF-06650808 3.0 mg/kg (Part 1) | PF-06650808 3.6 mg/kg (Part 1) | PF-06650808 4.68 mg/kg (Part 1) | PF-06650808 2.4 mg/kg (Part 2)
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 6 | 11 | 5 | 5 | 1 | 0
L/hr | NA (NA) — Summary statistics were not presented if fewer than 3 partipants had reportable parameter values. Individual participant values are 0.118 and 0.143 L/hr, respectively. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 0.0798 and 0.0808 L/hr, respectively. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 0.106 and 0.0703 L/hr, respectively. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 0.0894 and 0.124 L/hr, respectively. | 0.08368 (25) | 0.07545 (26) | 0.07924 (30) | 0.07517 (38) | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 0.0947 L/hr. |

12. Secondary Outcome: Volume of Distribution at Steady State (Vss) (Part 1 and Part 2)
Description: Vss was calculated as dose/(AUCinf × kel), where kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. Vss was only for PF-06650808 (ADC) and Cycle 1.
Time Frame: Pre-dose, 1, 4 and 24 hours post-dose, Days 4, 8 and 15 in Cycle 1
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | PF-06650808 0.2 mg/kg (Part 1) | PF-06650808 0.4 mg/kg (Part 1) | PF-06650808 0.8 mg/kg (Part 1) | PF-06650808 1.6 mg/kg (Part 1) | PF-06650808 2.0 mg/kg (Part 1) | PF-06650808 2.4 mg/kg (Part 1) | PF-06650808 3.0 mg/kg (Part 1) | PF-06650808 3.6 mg/kg (Part 1) | PF-06650808 4.68 mg/kg (Part 1) | PF-06650808 2.4 mg/kg (Part 2)
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 6 | 11 | 5 | 5 | 1 | 0
L | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values.Individual participant values are 3.43 and 3.45 L, respectively. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values.Individual participant values are 2.71 and 2.87 L, respectively. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values.Individual participant values are 3.51 and 2.20 L, respectively. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values.Individual participant values are 3.39 and 3.81 L, respectively. | 3.428 (26) | 3.232 (28) | 3.800 (30) | 3.481 (36) | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values.Individual participant values is 5.04. |

13. Secondary Outcome: Terminal Elimination Half-Life (t1/2) (Part 1 and Part 2)
Description: Terminal elimination half-life was defined as the time measured for the serum concentration to decrease by one half, and calculated as loge(2)/kel.
Time Frame: Pre-dose, 1, 4 and 24 hours post-dose, Days 4, 8 and 15 in Cycle 1 and Cycle 4
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | PF-06650808 0.2 mg/kg (Part 1) | PF-06650808 0.4 mg/kg (Part 1) | PF-06650808 0.8 mg/kg (Part 1) | PF-06650808 1.6 mg/kg (Part 1) | PF-06650808 2.0 mg/kg (Part 1) | PF-06650808 2.4 mg/kg (Part 1) | PF-06650808 3.0 mg/kg (Part 1) | PF-06650808 3.6 mg/kg (Part 1) | PF-06650808 4.68 mg/kg (Part 1) | PF-06650808 2.4 mg/kg (Part 2)
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 6 | 11 | 5 | 5 | 1 | 0
hr
  Serum PF-06650808 (ADC)_Cycle 1 | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 20.4 and 16.8 hr, respectively. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 23.5 and 24.9 hr, respectively. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 21.4 and 20.7 hr, respectively. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 27.2 and 20.1 hr, respectively. | 29.52 (5.2320) | 30.72 (5.0245) | 35.12 (4.1282) | 32.72 (5.1266) | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values is 40.8 hr. |
  Serum PF-06460005 (Total Antibody)_Cycle 1: number analyzed (Participants) | 1 | 2 | 1 | 2 | 6 | 10 | 5 | 5 | 1 | 0
  Serum PF-06460005 (Total Antibody)_Cycle 1 | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values is 19.1 hr. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 28.7 and 28.7 hr, respectively. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values is 28.4 hr. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 37.0 and 26.7 hr, respectively. | 33.62 (3.4487) | 40.93 (9.5650) | 49.06 (13.670) | 39.80 (9.2477) | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values is 61.1 hr. |
  Serum PF-06380101 (Unconjugated Payload)_Cycle 1: number analyzed (Participants) | 2 | 1 | 2 | 2 | 5 | 9 | 4 | 5 | 1 | 0
  Serum PF-06380101 (Unconjugated Payload)_Cycle 1 | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 45.2 and 26.5 hr, respectively. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values is 40.4 hr. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 50.3 and 39.9 hr, respectively. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 47.5 and 39.4 hr, respectively. | 53.06 (6.0260) | 53.11 (8.5249) | 59.18 (7.0486) | 53.52 (3.4434) | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values is 71.8 hr. |
  Serum PF-06650808 (ADC)_Cycle 4: number analyzed (Participants) | 0 | 1 | 1 | 2 | 4 | 4 | 0 | 2 | 0 | 0
  Serum PF-06650808 (ADC)_Cycle 4 |  | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values is 20.4 hr. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values is 18.5 hr. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 28.4 and 20.7 hr, respectively. | 28.50 (4.9349) | 30.33 (4.0991) |  | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 30.8 and 35.8 hr, respectively. |  |
  Serum PF-06460005 (Total Antibody)_Cycle 4: number analyzed (Participants) | 0 | 1 | 1 | 2 | 4 | 3 | 0 | 2 | 0 | 0
  Serum PF-06460005 (Total Antibody)_Cycle 4 |  | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values is 26.1 hr. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values is 24.6 hr. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 33.2 and 23.4 hr, respectively | 38.85 (3.7108) | 40.80 (2.5060) |  | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 41.8 and 59.2 hr, respectively |  |
  Serum PF-06380101 (Unconjugated Payload)_Cycle 4: number analyzed (Participants) | 0 | 1 | 1 | 2 | 4 | 4 | 0 | 2 | 0 | 0
  Serum PF-06380101 (Unconjugated Payload)_Cycle 4 |  | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values is 43.8 hr. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values is 38.8 hr. | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 45.7 and 49.2 hr, respectively. | 52.40 (7.9461) | 53.83 (6.5961) |  | NA (NA) — Summary statistics were not presented if fewer than 3 participants had reportable parameter values. Individual participant values are 48.7 and 61.5 hr, respectively. |  |

14. Secondary Outcome: Number of Participants With the Presence of Anti-PF-06650808 Antibodies (Part 1 and Part 2)
Description: Assays to assess for anti drug (anti PF-06650808) antibodies (ADA) were performed. Positive ADA: titer>=1.88.
Time Frame: 3 years
Population: The analysis population included all participants who received at least 1 dose of study medication and had at least 1 post-dose ADA measurements. The study was prematurely terminated prior to the start of dose expansion phase (Part 2).
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06650808 0.2 mg/kg (Part 1) | PF-06650808 0.8 mg/kg (Part 1) | PF-06650808 0.4 mg/kg (Part 1) | PF-06650808 1.6 mg/kg (Part 1) | PF-06650808 2.0 mg/kg (Part 1) | PF-06650808 2.4 mg/kg (Part 1) | PF-06650808 3.0 mg/kg (Part 1) | PF-06650808 3.6 mg/kg (Part 1) | PF-06650808 4.68 mg/kg (Part 1) | PF-06650808 2.4 mg/kg (Part 2)
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 7 | 11 | 6 | 6 | 2 | 0
Participants | 1 | 0 | 1 | 0 | 4 | 1 | 0 | 1 | 0 |

15. Secondary Outcome: Progression Free Survival and Overall Survival (Part 2)
Description: Progression Free Survival was defined as the time from Cycle 1 Day 1 (C1D1) to first documentation of disease progression or to death due to any cause, whichever occurs first. Overall survival was defined as the time from initial dose until death from any cause, and is measured in the intent to treat population.
Time Frame: 3 years
Population: The study was prematurely terminated prior to the start of dose expansion phase (Part 2).
Arm/Group | PF-06650808 2.4 mg/kg (Part 2)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- PF-06650808 0.2 mg/kg: PF-06650808 0.2 mg/kg was administered on Day 1 of each 21 day cycle per the DAI as an IV infusion over approximately 60 minutes.
- PF-06650808 0.4 mg/kg: PF-06650808 0.4 mg/kg was administered on Day 1 of each 21 day cycle per the DAI as an IV infusion over approximately 60 minutes.
- PF-06650808 0.8 mg/kg: PF-06650808 0.8 mg/kg was administered on Day 1 of each 21 day cycle per the DAI as an IV infusion over approximately 60 minutes.
- PF-06650808 1.6 mg/kg: PF-06650808 1.6 mg/kg was administered on Day 1 of each 21 day cycle per the DAI as an IV infusion over approximately 60 minutes.
- PF-06650808 2.0 mg/kg: PF-06650808 2.0 mg/kg was administered on Day 1 of each 21 day cycle per the DAI as an IV infusion over approximately 60 minutes.
- PF-06650808 2.4 mg/kg: PF-06650808 2.4 mg/kg was administered on Day 1 of each 21 day cycle per the DAI as an IV infusion over approximately 60 minutes.
- PF-06650808 3.0 mg/kg: PF-06650808 3.0 mg/kg was administered on Day 1 of each 21 day cycle per the DAI as an IV infusion over approximately 60 minutes.
- PF-06650808 3.6 mg/kg: PF-06650808 3.6 mg/kg was administered on Day 1 of each 21 day cycle per the DAI as an IV infusion over approximately 60 minutes.
- PF-06650808 4.68 mg/kg: PF-06650808 4.68 mg/kg was administered on Day 1 of each 21 day cycle per the DAI as an IV infusion over approximately 60 minutes.
Arm/Group | PF-06650808 0.2 mg/kg | PF-06650808 0.4 mg/kg | PF-06650808 0.8 mg/kg | PF-06650808 1.6 mg/kg | PF-06650808 2.0 mg/kg | PF-06650808 2.4 mg/kg | PF-06650808 3.0 mg/kg | PF-06650808 3.6 mg/kg | PF-06650808 4.68 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/2 | 1/7 | 1/11 | 0/6 | 0/6 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/2 | 1/7 | 3/11 | 3/6 | 3/6 | 2/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 2/2 | 2/2 | 7/7 | 11/11 | 6/6 | 6/6 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06650808 0.2 mg/kg (N=2) | PF-06650808 0.4 mg/kg (N=2) | PF-06650808 0.8 mg/kg (N=2) | PF-06650808 1.6 mg/kg (N=2) | PF-06650808 2.0 mg/kg (N=7) | PF-06650808 2.4 mg/kg (N=11) | PF-06650808 3.0 mg/kg (N=6) | PF-06650808 3.6 mg/kg (N=6) | PF-06650808 4.68 mg/kg (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06650808 0.2 mg/kg (N=2) | PF-06650808 0.4 mg/kg (N=2) | PF-06650808 0.8 mg/kg (N=2) | PF-06650808 1.6 mg/kg (N=2) | PF-06650808 2.0 mg/kg (N=7) | PF-06650808 2.4 mg/kg (N=11) | PF-06650808 3.0 mg/kg (N=6) | PF-06650808 3.6 mg/kg (N=6) | PF-06650808 4.68 mg/kg (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 2 | 3 | 0 | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foreign body sensation in eyes (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 3 | 2
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 4 | 1 | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 4 | 5 | 2 | 1 | 2
Rectal tenesmus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 5 | 2 | 0 | 0 | 2
Adverse drug reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 1 | 3 | 8 | 3 | 3 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Induration (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 2
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 0
Blood alkaline phosphatase (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood creatine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood parathyroid hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0
White blood cell count (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 4 | 2 | 1 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 4 | 5 | 6 | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 4 | 2 | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3 | 3 | 1 | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 4 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 4 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0
Nystagmus (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sedation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Menopausal symptoms (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 4 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 2 | 5 | 4 | 2 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 3 | 4 | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 2 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Systolic hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
The study was prematurely terminated as a business decision prior to the start of the dose expansion stage.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2014-05-07): https://cdn.clinicaltrials.gov/large-docs/05/NCT02129205/Prot_000.pdf
  • Statistical Analysis Plan (2014-11-17): https://cdn.clinicaltrials.gov/large-docs/05/NCT02129205/SAP_001.pdf